CLINICAL TRIAL: NCT07066657
Title: An Open-Label, Multi-Center, Dose Escalation, Confirmation, and Expansion Phase I Clinical Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of MRG007 (ARR-217) in Participants With Unresectable Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of MRG007 (ARR-217) in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lepu Biopharma Co., Ltd. (Industry)
Collaborators: ArriVent BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MRG007-001/ARR-217-101
Record Dates: First submitted 2025-06-26; First posted 2025-07-15 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced or Metastatic Solid Tumors; Colorectal Cancer; Gastric Cancer; Pancreatic Cancer
Keywords: MRG007; Advanced or Metastatic Solid Tumors; CDH17; ARR-217; ADC
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MRG007 (Experimental)
  Interventions: Drug: MRG007

INTERVENTIONS:
Drug: MRG007 — MRG007 will be administrated as specified in the protocol.
  Other Names: ARR-217

SUMMARY:
This is an open-label, multi-center, phase I study to evaluate the safety, tolerability, efficacy, and pharmacokinetics of MRG007 (ARR-217) in patients with unresectable locally advanced or metastatic solid tumors.

ELIGIBILITY:
1. Willing to sign the informed consent form and follow the requirements specified in the protocol.
2. Life expectancy ≥ 3 months.
3. Tumor specimen available for CDH17 testing, or agree to biopsy at baseline.
4. Patients with histologically and cytologically confirmed advanced or metastatic solid tumor who have failed or intolerant to standard therapy, or without alternative standard therapy.
5. Patients must have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
6. The score of ECOG for performance status is 0 or 1.
7. Organ functions and coagulation function must meet the basic requirements.
8. Patients with childbearing potential must use effective contraception during the treatment and for 6 months after the last dose of treatment.

Exclusion Criteria:

1. Patients with more than one cancer.
2. Received CDH17-targeting anti-tumor therapy; received other investigational product, systemic corticosteroids or surgery for major organs within 4 weeks prior to the first dose; received anti-tumor therapy within 3 weeks or within 5 half-lives prior to the first dose, whichever is shorter; received radiotherapy within 2 weeks prior to the first dose; received potent CYP3A4 inducers or inhibitors within 2 weeks prior to the first dose or 5 half-lives of investigational product, whichever is longer.
3. ≥Grade 2 toxic reaction or abnormal value of laboratory test caused by previous anti-tumor treatment
4. Symptomatic Central nervous system and/or meninges metastasis.
5. History of severe cardiovascular diseases
6. Cerebrovascular accident, pulmonary embolism, or deep venous thrombosis within 3 months prior to the first dose, implantable venous infusion port or catheter-related thrombosis, or superficial venous thrombosis
7. History of previous or combined interstitial pneumonia, current interstitial pneumonia, or suspected interstitial pneumonia that cannot be ruled out through imaging during screening, severe chronic obstructive pulmonary disease with respiratory failure, severe pulmonary dysfunction, symptomatic bronchospasm, etc.
8. Poorly controlled pleural, peritoneal, and pelvic effusion, or combined pericardial effusion
9. Infection of active hepatitis B, active hepatitis C, or HIV
10. Uncontrolled active bacterial, viral, fungal, rickettsial, or parasitic infections requiring intravenous anti-infection therapy within 2 weeks prior to the first study treatment
11. Known allergic reactions to any component of MRG007, or known Grade≥3 allergic reactions to other prior anti-CDH17 (including investigational) or other monoclonal antibody.
12. Other situations that are not suitable to participate a clinical trial per investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) - Phase Ia | Baseline to Day 21 of the first treatment cycle
Serious Adverse Events (SAEs) | Baseline to 30 days after the last dose of study treatment
  Adverse events that are fatal, life-threatening, or result in hospitalization or prolonged hospitalization, persistent or significant disability/incapacity/substantial disruption of the ability to lead a normal life, congenital anomaly/birth defect or major medical events or reactions
Treatment-Emergent Adverse Event (TEAE) | Baseline to 30 days after the last dose of study treatment
  AEs that occur or worsen on or after the first dose of study treatment
Treatment-Related Adverse Event | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial is considered related to the study drug.
Objective Response Rate (ORR) as assessed by investigator - Phase Ib | Baseline to study completion (up to 24 months)
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed according to RECIST v1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) - Phase Ia | Baseline to study completion (up to 24 months)
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed according to RECIST v1.1.
Disease Control Rate (DCR) | Baseline to study completion (up to 24 months)
  DCR is defined as the proportion of subjects achieving CR, PR, and stable disease (SD) after treatment.
Duration of Response (DOR) | Baseline to study completion (up to 24 months)
  The time interval between the date of the earliest qualifying response and the date of disease progression or death for any cause, whichever occurs earlier.
Progression Free Survival (PFS) as assessed by investigator | Baseline to study completion (up to 24 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Overall Survival (OS) | Baseline to study completion (up to 24 months)
  OS is defined as the duration from the start of treatment to death of any cause.
Incidence of anti-drug antibody (ADA) | Baseline to 30 days after the last dose.
  The proportion of patients with positive ADA results.
Incidence of neutralizing antibody (NAb) | Baseline to 30 days after the last dose.
  The proportion of patients with positive NAb results.
Tmax | Baseline to 30 days after the last dose of study treatment
  Time to reach the maximum blood concentration
Cmax | Baseline to 30 days after the last dose of study treatment
  Maximum observed blood concentration
AUC0-t | Baseline to 30 days after the last dose of study treatment
  Area under the blood concentration-time curve from time 0 to the time of last quantifiable concentration

CONTACTS AND LOCATIONS:
Locations (15):
- United States (10):
  - ULCA, Los Angeles, California
  - UCSF, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Sarah Cannon Research Institute, Denver, Colorado
  - Sarah Cannon Research Institute, Sarasota, Florida
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Dallas, Irving, Texas
  - NEXT Virginia, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- China (5):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No